CLINICAL TRIAL: NCT05688488
Title: Clinical Study of Curcumin in Preventing Postoperative Adhesion of Bilateral Vocal Cords
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022011-1
Record Dates: First submitted 2022-12-28; First posted 2023-01-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-01

CONDITIONS: Glottic Web of Larynx; Laryngeal Stenosis; Glottic Carcinoma; Laryngeal Leucoplakia; Laryngeal Polyp; Laryngeal Papilloma
Keywords: Curcumin
MeSH Terms: conditions — Laryngostenosis; Laryngeal papillomatosis | interventions — Curcumin; Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin (Experimental)
  Interventions: Drug: Curcumin
- Mitomycin (Active Comparator)
  Interventions: Drug: Mitomycin-C

INTERVENTIONS:
Drug: Curcumin — Curcumin was applied to both wound sites of bilateral vocal cords. After evenly applied, gently massage the applied site for 3-5 minutes until the drug was fully absorbed.
  Arms: Curcumin
Drug: Mitomycin-C — Mitomycin-C was applied to both wound sites of bilateral vocal cords. After evenly applied, gently massage the applied site for 3-5 minutes until the drug was fully absorbed.
  Arms: Mitomycin

SUMMARY:
To provide a novel therapy idea and method to solve the clinical problem of postoperative adhesion of bilateral vocal cords, patients enrolled in this study will be applied with curcumin on both wound sites of bilateral vocal cords after the surgery on the bilateral vocal cord endoscopically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral vocal cord diseases who are going to undergo resection of bilateral vocal cord lesions endoscopically.
2. Patients with bilateral vocal cord adhesion who are going to undergo incision of bilateral vocal cord adhesion endoscopically.

Exclusion Criteria:

1. Patients with other laryngeal diseases.
2. Patients with cardiac and pulmonary insufficiency.
3. Patients unable to cooperate with the follow-up on time after surgery.
4. Patients who refuse to sign the informed consent after notification.
5. Patients who have a severe allergic disease or allergic history to a variety of drugs.
6. Other circumstances that are not appropriate to be included in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with laryngeal web formation as assessed by videolaryngoscope | 1 year postsurgery
  All participants received the videolaryngoscope every month post-surgery, and a laryngeal web is defined as a visible adhesion whose length reached 1 mm or greater.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided